CLINICAL TRIAL: NCT02034617
Title: Evaluation of a Parent-Infant Interaction Model in the Neonatal Intensive Care
Brief Title: Evaluation of a Parent-Infant Interaction Model
Acronym: LiMoNid
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Linkoeping University (Other Government)
Responsible Party: Principal Investigator, Evalotte Morelius, Professor, Linkoeping University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: LinkoepingU
Record Dates: First submitted 2013-12-19; First posted 2014-01-13 (Estimated); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Premature Birth
Keywords: Cognition; Family nursing; Infant, premature; Object attachment; Stress, physiological; Stress, psychological
MeSH Terms: conditions — Premature Birth; Stress, Psychological

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard care (No Intervention): The family receive standard care when enrolled in the Neonatal intensive care unit
- Observation (Experimental): The family receive standard care when enrolled in the Neonatal intensive care unit and are also included in an observational program called LiMoNid.
  Interventions: Behavioral: LiMoNid

INTERVENTIONS:
Behavioral: LiMoNid — One LiMoNid observation will be performed on day 1-3 post birth, one in time of discharge, and one in the home when the infant has reached 40 weeks (+/- 2 week). All observations are performed in presence of and in collaboration with the parents with the outspoken aim to guide the parents to learn how to read and respond to their infant' signals
  Arms: Observation

SUMMARY:
When becoming a parent of a preterm infant there is an increased risk of stress. There are a number of studies showing that parental stress has a negative impact on their engagement with their child. Other studies, on the other hand, show that different intervention programs with the aim to strengthen the relationship can decrease parental stress and hence affect the parent-infant interaction in a positive way. Structured intervention programs for preterm infants have also been successful in improving the infants' cognitive functions.

The investigators have developed a program with the aim to strengthen the parent-infant interaction for late preterm infants. The observational program is called LiMoNid. Our hypothesis is that LiMoNid will strengthen the parents' own parental abilities and give them a deeper understanding of their child. They will hopefully develop more skills on how to communicate with their child; to see, interpret, understand and approach the child, which can lead to an improved parent-child interaction. Parental stress may also be reduced by increased understanding and control. Regarding the child itself, we hypothesize that the psychological development will be affected depending on the communication with the caregiver and depending on the support it has received in expressing its feelings and needs. The emotional regulation should be strengthened by such an intervention.

The aim is to study if LiMoNid can have an impact on cognition, stress, parent-child interaction.

DETAILED DESCRIPTION:
The Design is a randomised controlled study in two groups; intervention group versus standard care. Parents who meet the inclusion criteria are given oral and written information about the study aim and procedure and are asked for participation. If the parents consent they will be randomised to one of two groups. Follow-ups will be conducted at 1 month, 4 months, 10-12 months corrected age and when the child is 4 years.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants born 30-36 weeks gestational age without known major malformations or complications
* Families living in the county of Ostergotland, Sweden
* Swedish speaking parents
* Single or duplex birth

Exclusion Criteria:

* Complications encountered during hospital stay that are known to affect cognition

Max Age: 96 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Cognitive abilities | 11 months
  Bayley Scales of Infant Development

SECONDARY OUTCOMES:
Stress reactivity | 1 month
  Salivary cortisol reactivity in relation to bath

OTHER OUTCOMES:
Parent-child interaction | 1 month
  Ainsworth sensitivity scale
Stress reactivity | 4 months
  Salivary cortisol reactivity in relation to still-face
Parent-child interaction | 4 months
  Still-face and Ainsworth sensitivity scale
Parental stress | 1 month
  Edinburgh Post Depression Scale (EPDS) and State-Trait and Anxiety Inventory, short version (STAI)
Parental stress | 4 months
  Edinburgh Post Depression Scale (EPDS), State-Trait and Anxiety Inventory, short version (STAI) and Swedish Parenthood Stress Questionnaire (SPSQ)
Parent-child interaction | 11 months
  Infant Parent Social Interaction (IPSIC) and Attachment Story Stems
Stress reactivity | 11 months
  Salivary cortisol reactivity in relation to a standardized play-situation, Infant Parent Social Interaction (IPSIC)
Parental stress | 11 months
  State-Trait and Anxiety Inventory, short version (STAI) and Swedish Parenthood Stress Questionnaire (SPSQ)
Emotions | 11 months
  Ages and Stages Questionnaire: Social and emotional (ASQ-SE)
Cognitive abilities | 4 years
  Wechsler Preschool and Primary Scale of Intelligence (WPPSI-III)
Parental stress | 4 years
  State-Trait and Anxiety Inventory, short version (STAI)
Parental style | 4 years
  Parenting Scale (PS)
Emotions | 4 months
  Ages and Stages Questionnaire: Social and emotional (ASQ-SE)
Emotions | 4 years
  Ages and Stages Questionnaire: Social and emotional (ASQ-SE) and Emotion Regulation Questionnaire for Children

CONTACTS AND LOCATIONS:
Overall Officials: Evalotte Morelius, PhD, Principal Investigator — Linkoeping University
Locations (1):
- Linkoping University Hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Helmer CS, Thornberg UB, Abrahamsson T, Morelius E. Mothers' experiences of a new early collaborative intervention, the EACI, in the neonatal period: A qualitative study. J Clin Nurs. 2023 Jun;32(11-12):2892-2902. doi: 10.1111/jocn.16412. Epub 2022 Jun 14. PMID 35702001
- [Result] Helmer CS, Thornberg UB, Morelius E. An Early Collaborative Intervention Focusing on Parent-Infant Interaction in the Neonatal Period. A Descriptive Study of the Developmental Framework. Int J Environ Res Public Health. 2021 Jun 21;18(12):6656. doi: 10.3390/ijerph18126656. PMID 34205660
- [Derived] Birberg Thornberg U, Koch FS, Helmer CS, Tell J, Nyberg E, Abrahamsson T, Morelius E. Moderate-To-Late Preterm Infants Benefit From the Early Collaborative Intervention: Primary Outcomes of an RCT. Acta Paediatr. 2025 Nov;114(11):2838-2846. doi: 10.1111/apa.70173. Epub 2025 Jun 13. PMID 40511708